CLINICAL TRIAL: NCT01653769
Title: CoSeal for Hemostasis of Aortic Anastomoses: A Propensity-Matched Cohort Study
Brief Title: CoSeal for Hemostasis of Aortic Anastamoses
Status: Completed | Type: Observational
Sponsor: Michael Reardon, MD (Other)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor-Investigator, Michael Reardon, MD, Sponsor-Investigator/Principal Investigator, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Other Study IDs: Pro00007251; IRB(2)0312-0064 (Other: TMHRI IRB); BS11-000639 (Other: Other ID)
Record Dates: First submitted 2012-07-02; First posted 2012-07-31 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Surgical Bleeding; Aneurysms; Aortic Dissection
Keywords: CoSeal; Surgical bleeding; hemostasis; Aortic anastamoses; bleeding; Cardiac surgery; Aneurysms; Aortic Dissection
MeSH Terms: conditions — Aneurysm; Aortic Dissection; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: None Retained — Time perspective is both retrospective and prospective.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Surgery on the aorta can be associated with significant blood loss. Most commonly this is due to bleeding at the site of aortic anastomosis. Surgical bleeding is associated with significant morbidity.

One way to prevent bleeding is to use a special glue (sealant) after performing large connections on the aorta. The goal of this study is to compare the different methods surgeons use to stop/prevent bleeding.

The study team will collect medical information about patients before, during, and after surgery on their aortas, including the methods used to prevent bleeding. This information may help doctors improve the way that they care for these patients.

DETAILED DESCRIPTION:
Bleeding is a major complication of cardiac surgery, and a significant cause of morbidity and mortality [1-4]. Hemostasis can be challenging during complex cardiac surgery, particularly due to friability of the tissue, coagulopathy, poor visualization of the surgical field, and limited accessibility to bleeding sites [5]. Failure to achieve and maintain hemostasis and reinforce fragile tissue may result in additional bleeding, which can further reduce visualization, increase operative blood loss, lengthen surgery, increase the use of blood products, and contribute to postoperative complications and reoperation [1-4].

Postoperative bleeding is a significant concern in cardio-thoracic surgery. Bleeding, either intraoperative or postoperative, has been associated with extended in-hospital length of stay, reoperations, severe morbidity and death [12]. In addition to surgical technique, a variety of therapeutic agents are available to assist in hemostasis. Surgical sealants are used to prevent suture line bleeding when ligation or conventional methods are ineffective or impractical [13]. CoSeal® Surgical Sealant (CoSeal®, Baxter, Westlake Village, CA) is a synthetic polyethylene glycol (PEG) polymer [11, 13]. The polymers cross-link with proteins in the tissue and begin to gel in approximately 5 seconds and set within 60 seconds, forming a strong, flexible, clear, degradable hydrogel that adheres to both tissue and synthetic graft surfaces [11, 13-14]. A secure seal is maintained through covalent tissue bonds even under high pressures in vessels, such as the aorta [15]. The gel is completely resorbed within 30 days [14].

ELIGIBILITY:
Inclusion Criteria:

* The study will include all patients undergoing cardio-thoracic surgery requiring a large aortic anastomosis.

Exclusion Criteria:

* Patients with severe preoperative coagulopathy, connective tissue disorders and disseminated intravascular coagulopathy (DIC) will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects for this study will be selected from patients undergoing cardio-thoracic surgery requiring a large aortic anastomosis. Both the retrospective and prospective study components will review the data of all procedures requiring a large aortic anastomosis in order to compare those in which CoSeal® was used versus other materials/techniques.
  For the retrospective arm of the study, pre-existing data will be collected from the patient's medical records under a HIPAA Waiver of Authorization. For the prospective arm of the study, patients will provide consent to collect their data.
  Approximately 150 patients will be enrolled in this study. Specifically, consecutive potential subjects will be evaluated for participation in this study according to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-06; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
reduction in intra- and post-operative bleeding for procedures using CoSeal for hemostasis | from day of surgery to 15-30 days after discharge
  estimated blood loss/chest drain output; blood product requirement during surgery; re-operation for bleeding

SECONDARY OUTCOMES:
decrease length of stay | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  length of stay (LOS) in ICU, LOS in-hospital (admission to discharge); day of surgery to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Michael Reardon, MD, Principal Investigator — The Methodist Hospital Department of Cardiovascular Surgery
Locations (1):
- The Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share available data.